CLINICAL TRIAL: NCT00566137
Title: Sleep Disturbances and Pulmonary Artery/Aorta Diameter in Scleroderma Patient
Acronym: Scleroderma
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: ARUNABH TALWAR MD, NORTH SHORE- LONG ISLAND HEALTH SYSTEM
Other Study IDs: 06-08-018; NS-LIJHS IRB #06-08-018
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Scleroderma; Pulmonary Hypertension
Keywords: Scleroderma; Pulmonary Hypertension
MeSH Terms: conditions — Scleroderma, Diffuse; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine sleep disturbance, pulmonary function test, 6 minute walk, echocardiogram abnormality, arterial blood gas, ventilation/perfusion scan of the chest in Scleroderma patient with Pulmonary Hypertension.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* Patient must have Scleroderma

Exclusion Criteria:

* Patients who do not have Scleroderma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males, Females and Minorities
  Age range of subjects 18-75 years old
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-02; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arunabh Talwar, MD, Principal Investigator — Northwell Health